CLINICAL TRIAL: NCT00918515
Title: A Phase I, Single-Centre, Open Label Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intravenous AZD3043 After Single Ascending Doses in Healthy Male Volunteers
Brief Title: Study to Assess the Safety, Tolerability and Pharmacokinetics and Pharmacodynamics of AZD3043
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Stephen Kanes, Medical Science Director, AstraZeneca Pharmaceuticals US
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0510C00001; 2007-003474-26
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2009-08

CONDITIONS: Healthy
Keywords: Sedation; Anaesthesia; Safety; tolerability; pharmacokinetics; pharmacodynamics; healthy male volunteers
MeSH Terms: interventions — AZD-3043

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD3043 (Experimental): Intravenous solution
  Interventions: Drug: AZD3043

INTERVENTIONS:
Drug: AZD3043 — intravenous solution given once as intravenous infusion over 30 minutes

SUMMARY:
This is a Phase I, single centre, open label study to assess the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics of intravenous AZD3043 after single ascending doses in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 18 to 45 years with suitable veins for cannulation or repeated venepuncture
* Pre-dose assessment judged without remarks by the investigator
* Have a Body Mass Index (BMI) between 19 and 30 kg/m2 and weight at least 50kg and no more than 100kg

Exclusion Criteria:

* After adequate time (at least 15 minutes) of rest in supine position, abnormal vital signs defined as any of the following:·
* Systolic blood pressure (BP) >140 mm Hg.·
* Diastolic BP >90 mm Hg.
* Heart rate <=55 or >85 beats per minute
* Subjects with compromised airway or respiratory function as evidenced by the presence of Class 3 or 4 Airway, Sleep Apnoea, Neck circumference > 16.5 inches (42 cm), Asthma, Active or recent (2 weeks) respiratory infection, or known chronic respiratory infection, or known chronic respirator
* Lack of a normal phenotype for butyrylcholinesterase (pseudo-cholinesterase)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2009-05; Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Assessment of Vital signs data, heart rate, electrocardiogram (ECG) | The measure will be taken between -20 to 150 min relative to start of administration of AZD3043.
Respiratory signs data (SpO2, EtCO2, PaO2, blood gases, respiratory frequency, volume and pattern, occurrence of apnoea; | The measure will be taken between -20 to 150 min relative to start of administration of AZD3043.

SECONDARY OUTCOMES:
PK parameters for AZD3043: Cmax (Css), AUClast, AUC, lz, t½lz, CL, Vc, Vss, Vz, tlast and mean residence time in arterial and venous plasma. | Arterial: Predose, 2, 5, 15, 29, 31, 32, 35, 37, 40, 45, 60, 75, 90, 150 min postdose. Venous: Predose, 2, 5, 15, 29, 31, 32, 35, 37, 40, 45, 60, 75, 90, 150, 270 min, 8h, 24h postdose.
PK parameters for the metabolite (THRX 108893): Cmax (Css), AUClast, AUC, tmax, tlast, lz and t½lz in venous plasma | 29 min, 45 min and 150 min post dose

CONTACTS AND LOCATIONS:
Overall Officials: Johan Wemer, Study Chair — AstraZeneca R&D Södertälje; Sigridur Kalman, Principal Investigator — Department of Clinical Science Intervention and technology, CLINTECThe department of Anaesthosiology and Intensive care, Karolinska University hospital, Huddinge,141 86 Stockholm, Sweden
Locations (1):
- Research Site, Stockholm, Sweden